CLINICAL TRIAL: NCT01967680
Title: Non-sedation Versus Sedation With a Daily Wake-up Trial in Critically Ill Patients Receiving Mechanical Ventilation. The NONSEDA-trial. An Investigator-initiated, Randomised, Clinical, Parallel-group, Multinational, Superiority Trial
Brief Title: Non-sedation Versus Sedation With a Daily Wake-up Trial in Critically Ill Patients Receiving Mechanical Ventilation
Acronym: NONSEDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palle Toft (Other)
Collaborators: The Danish Medical Research Council (Other); Aase and Ejnar Danielsens Foundation (Other)
Responsible Party: Sponsor-Investigator, Palle Toft, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-20130025
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Critical Illness; Respiration, Artificial
MeSH Terms: conditions — Critical Illness; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sedation with daily wake-up trial (Active Comparator): The control group is sedated with continuous infusion to Ramsay score 3-4. During daytime, the patient is awakened as the intravenous infusion of sedatives is discontinued. After a successful wake-up, the infusion of sedative is resumed, starting on half of the pre-wake-up dose. If the patient becomes uncomfortable or agitated during the awakening, sedation is resumed, again starting with half the dosage. The infusion of sedatives is then adjusted to Ramsey score 3-4.
  Interventions: Procedure: Controlgroup, sedation with daily wake-up trial
- Non-sedation (Experimental): This group will not receive sedatives. Patients are thoroughly and repeatedly informed by the staff of where they are, what have happened, and what type of treatment they are going to receive.
  Participants in the non-sedated group are awake and have a natural sleep rhythm. In case these patients develop and outward delirium, it is necessary to have a nurse or other caregiver at the bedside in order to calm the patient. Patients with delirium are treated with haloperidol according to the U.S. guidelines, 2002 and the Danish national guidelines.
  If, despite these measures, it is necessary to sedate an agitated patient more than twice, or where sedation might be necessary to ensure sufficient oxygenation or prone position, the patient is sedated and treated like the control-group. Every day during the wake-up trial it is evaluated whether the patient is able to continue the intervention of non-sedation.
  Interventions: Procedure: Non-sedation for intubated, mechanically ventilated patients

INTERVENTIONS:
Procedure: Non-sedation for intubated, mechanically ventilated patients
  Arms: Non-sedation
Procedure: Controlgroup, sedation with daily wake-up trial
  Arms: Sedation with daily wake-up trial

SUMMARY:
Background: Every year 30,000 Danish patients are admitted to Intensive Care Units (ICU), accounting for 2-3% of all patients in hospital and 30% of the yearly hospital expenditure. The mortality in the ICU is 12.7 % and the 30-day mortality is 21.2 % according to the national Danish Intensive Care Database. Through many years, the standard care has been to use continuous sedation of critically ill patients during me-chanical ventilation. However, recent research indicates that it is beneficial to reduce the sedation level in these patients. A randomised trial found that continuous sedation with a daily wake-up trial compared to continuous sedation reduced the time on me-chanical ventilation and the length of stay in the intensive care unit. Further, a ran-domised trial comparing continuous sedation with a daily wake-up trial to no sedation found that patients in the non-sedated group needed mechanical ventilation for a shorter time and had a shorter length of stay in the ICU and in the hospital. The trial also indicated a beneficial effect on mortality, however the trial was not a priori de-signed or powered with respect to mortality. No randomised trial has been published comparing sedation with no sedation, a priori powered to have all-cause mortality as primary outcome.

Objective: To assess the benefits and harms of non-sedation versus sedation with a daily wake-up trial in critically ill patients in ICU.

Design: The NONSEDA trial is an investigator-initiated, randomised, clinical, parallel-group, multinational, superiority trial designed to include 700 patients from at least six ICUs in Denmark, Norway and Sweden.

Inclusion criteria: Mechanically ventilated patients with expected duration of me-chanical ventilation > 24 hours.

Exclusion criteria: non-intubated patients, patients with severe head trauma, coma at admission or status epilepticus, patients treated with therapeutic hypothermia, patients with PaO2/FiO2<9 where sedation might be necessary to ensure sufficient oxygenation or place the patient in prone position.

Experimental intervention: Non-sedation supplemented with pain management during mechanical ventilation.

Control intervention: Sedation with a daily wake-up trial.

The primary hypothesis is that non-sedation compared to sedation and a daily wake-up trial will reduce mortality.

The secondary hypotheses are that non-sedation compared to sedation and a daily wake-up trial will:

* Reduce the incidence of a composite outcome of death, acute myocardial in-farction (AMI), stroke, pulmonary embolism and other thromboembolic events.
* Reduce the number of organ failures.
* Increase the days alive without mechanical ventilation.
* Increase the days alive outside the ICU.
* Increase the days alive outside the hospital.

Outcomes: The primary outcome is all-cause mortality at 90 days. Secondary out-comes are time to death in the trial period, the frequency of the trombo-embolic com-plications, acute renal failure, days alive without mechanical ventilation, days alive outside the ICU and hospital. Explorative outcomes are mortality at 28 days, organ failure and coma-free, delirium-free days.

Trial size: The investigators will include 700 participants (2 x 350) in order to detect or reject 25% relative risk reduction in mortality with a type I error risk of 5% and a type II error risk of 20% (power at 80%).

ELIGIBILITY:
Inclusion Criteria:

Endotracheally intubated Expected time on ventilator > 24 h. Age ≥ 18 years Informed consent

Exclusion Criteria:

Severe head trauma where therapeutic coma is indicated Therapeutic hypothermia where therapeutic coma is indicated Status epilepticus where therapeutic coma is indicated Patient has participated in the study before Patient is transferred from another ICU with length of stay > 48 hours Patient is comatose at admission PaO2/FiO2 ≤ 9, if sedation is necessary for oxygenation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Mortality | 90 days
  All cause mortality at 90 days after randomization

SECONDARY OUTCOMES:
Days until death | 1 year
  Days until death throughout the total observation period
Cardiovascular event | 90 days
  Proportion of participants with a major cardiovascular outcome (acute myocardial infarction, cerebral infarction, cerebral hemorrhage, pulmonary embolus, deep vein thrombosis, other thrombo-embolic event) at 90 days after randomization.
Coma and deliriumfree days | 28 days
  Number of coma- and delirium-free days (defined as RASS ≥ 3 and no positive CAM-ICU scorings the particular day) within 28 days from randomization
RIFLE-score | 28 days
  Highest Rifle-score within 28 days from randomization (Rifle-categories: Rifle-R: Increase in serum creatinine x 1.5 from baseline OR urine output < 0.5 mL/kg/hr x 6 h.
  Rifle-I: Increase in serum creatinine x 2 from baseline OR urine output < 0.5 mL/kg/hr x 12 h.
  Rifle-F: Increase in serum creatinine x 3 from baseline OR urine output < 0.3 mL/kg/hr x 24h OR creatinine ≥ 350μmol/L with acute rise ≥ 44 μmol/L in < 24h)
Days until discharge | 28 days
  Days until discharge from ICU (within 28 days from randomization).
Days until the participant is without mechanical ventilation | 28 days
  Days until the participant is without mechanical ventilation (within 28 days from randomization).

OTHER OUTCOMES:
Mortality | 28 days
  All cause mortality at 28 days after randomisation.
Discharge fro ICU | 90 days
  Days until discharge from the intensive care unit (within 90 days from randomization)
End of mechanical ventilation | 90 days
  Days until the participant is without without mechanical ventilation (within 90 days from randomization)
Discharge from hospital | 90 days
  Days until discharge from the hospital (within 90 days from randomization).
Number of organ failures | ICU-admission
  Organ failure when the patient is discharged from the ICU.
Accidental extubation | ICU-admission
  Number of accidental extubations requiring re-intubation within 1 hour
Accidental removal of cental venous line | ICU-admission
  Number of accidental removals of central venous lines, requiring re-insertion within 4 hours
Oxygenation | During ventilator treatment
  Worst oxygenation status measured by
  * highest fraction of oxygen in inspired air (FiO2)
  * worst paO2/FiO2-ratio registered daily
1-year survival | 1 year from randomisation
  Number of patients alive 1 year after randomisation in each group

CONTACTS AND LOCATIONS:
Overall Officials: Palle Toft, Professor, Study Chair — Odense University Hospital; Hanne Tanghus Olsen, MD, Principal Investigator — Svendborg Hospital; Helene K Nedergaard, MD, Principal Investigator — Kolding Sygehus; Thomas Stroem, Postdoc, Principal Investigator — Odense University Hospital
Locations (8):
- Denmark (5):
  - Sydvestjysk Sygehus, Esbjerg, Region Syddanmark
  - AArhus university Hospital, Noerrebrogade, Aarhus
  - Kolding Hospital, Kolding
  - Odense University Hospital, Odense
  - Svendborg Hospital, Svendborg
- Norway (2):
  - University Hospital of North Norway, Tromsø
  - Vestfold Hospital, Tønsberg
- Linkjøbing University Hospital, Linköping, Sweden

REFERENCES:
- [Background] Strom T, Martinussen T, Toft P. A protocol of no sedation for critically ill patients receiving mechanical ventilation: a randomised trial. Lancet. 2010 Feb 6;375(9713):475-80. doi: 10.1016/S0140-6736(09)62072-9. Epub 2010 Jan 29. PMID 20116842
- [Derived] Oxlund J, Knudsen T, Strom T, Lauridsen JT, Jennum PJ, Toft P. Serum melatonin concentration in critically ill patients randomized to sedation or non-sedation. Ann Intensive Care. 2021 Mar 6;11(1):40. doi: 10.1186/s13613-021-00829-1. PMID 33677695
- [Derived] Olsen HT, Nedergaard HK, Strom T, Oxlund J, Wian KA, Ytrebo LM, Kroken BA, Chew M, Korkmaz S, Lauridsen JT, Toft P. Nonsedation or Light Sedation in Critically Ill, Mechanically Ventilated Patients. N Engl J Med. 2020 Mar 19;382(12):1103-1111. doi: 10.1056/NEJMoa1906759. Epub 2020 Feb 16. PMID 32068366